CLINICAL TRIAL: NCT06870799
Title: Randomized Controlled Trial Comparing Closed Face Masks vs Surface Guided Radiation Therapy for Head and Neck Radiotherapy
Brief Title: Comparing Closed Face Masks vs Surface Guided Radiation Therapy for Head and Neck Radiotherapy
Acronym: NoMask
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAO 24-019; 2025-D0007 (Other: BASEC)
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancers
Keywords: head and neck cancer; face mask; surface guidance; radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Closed Mask followed by No Mask (Other): The first half of the treatment is delivered with a face mask, the second half is delivered without mask using surface guidance only
  Interventions: Device: Surface guided radiation therapy; Device: Closed face mask
- No Mask followed by Closed Mask (Other): The first half of the treatment is delivered without mask using surface guidance only, the second half is delivered with a face mask
  Interventions: Device: Surface guided radiation therapy; Device: Closed face mask

INTERVENTIONS:
Device: Surface guided radiation therapy — Radiation therapy will be delivered using no immobilization mask, but a surface guided system with infrared light
Device: Closed face mask — Radiotherapy with closed face mask for immobilization

SUMMARY:
At present, open-face masks are used only in patients with claustrophobic anxiety, while all other patients are still immobilized with closed masks, thereby overlooking the need for improvement in patient comfort. Closed face masks in patients undergoing head and neck irradiation have never been compared to no masks in the setting of a randomized clinical trial, but only in feasibility trials. A randomized clinical trial may establish the role of no masks in terms of patient comfort, preference and setup accuracy in all patients.

DETAILED DESCRIPTION:
Once eligibility has been confirmed and upon randomization, patients will begin treatment either with an immobilization mask (A) or no mask (B). One individual immobilization mask and AccuForm cushion will be fabricated for every single patient. All positioning setup information used for subsequent treatment sessions will be documented. One simulation CT/MRI will be acquired and one treatment plan for each setup. After image acquisition, the mask will be removed and stored for treatment. After the simulation, the patients will be asked to fill out a questionnaire evaluating their comfort/anxiety/pain in regards to the setup as a baseline assessment. The patients will be treated with 6 MV from a linear accelerator (Truebeam, Varian Medical Systems, Palo Alto, CA). Dose prescription and treatment planning objectives of the individual patient will be defined by the standard treatment protocol depending on the patient's disease and treatment intention. Before each treatment session, the patient will be positioned on the treatment couch with the designated immobilization material. Conebeam-CT (CBCT) images will be acquired followed by automatic/manual setup correction compared to simulation CT/MRI; a CBCT image will be acquired after the treatment session once a week and at the first three fractions with mask and no mask. The CBCT procedure is a part of the standard treatment protocol for head-and-neck irradiation. Data on CBCT imaging in the form of translational and rotational shifts will be used to measure and compare setup uncertainties (inter-fraction and intra-fraction accuracy) between the two arms. In the no mask arm, Align RT® (Vision RT Ltd., UK) an SGRT system will be used in addition to CBCT imaging, to evaluate translational and rotational motions during treatment and for initial set up and also Gate during treatment. The SGRT system will not be used in patients with immobilization masks on. On the first day of treatment and weekly thereafter (immediately after treatment), the patients will be asked to fill out the same questionnaire as in Simulation for a comfort/anxiety/pain evaluation. As standard practice, patients typically receive another CT simulation during the second half of their treatment, to allow for adjustments to their radiation plan. This is typically due to factors such as weight loss, swelling, tumour or anatomical changes. If necessary, a new mask is also created to account for such changes. This workflow will apply to this study and participants. At the very last treatment session, they will answer the question on their mask or no mask preference.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before any trial specific procedures;
* Indication for head and neck radiotherapy irrespective of tumor type;
* Age: ≥ 18 years old;
* Karnofsky performance status ≥70;
* Patients who are willing and able to comply with scheduled visits, treatment, and other trial procedures.

Exclusion Criteria:

* Prior head and neck irradiation;
* Women who are pregnant or breast feeding;
* Intention to become pregnant during the course of the trial;
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases;
* Known or suspected non-compliance, drug or alcohol abuse;
* Inability to follow the procedures of the trial, e.g. due to language problems of the participant;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* One of the following Tumor Types: Nasopharynx, Sinunasal, patients with CTV within 5 mm of eyes or spinal cord.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Patient discomfort, anxiety and pain | weekly from enrollment to end of treatment up to 7 weeks
  Patients are asked to fill in a short questionnaire to rate their discomfort, anxiety and pain on a visual analogue scale ranging from 0 (=none) to 10 (=extreme)
overall preference | once at end of treatment (max. 7 weeks)
  patients are asked to answer the question which treatment modality they preferred (with mask or without mask)

SECONDARY OUTCOMES:
Setup uncertainties | during treatment before every treatment fraction, 5-6 times per week up to 7 weeks
  inter-fraction accuracy is measured with CBCT imaging
intra-fraction accuracy | during treatment before every treatment fraction, 5-6 times per week up to 7 weeks
  intra-fraction accuracy is measured with planar CBCT imaging and an optic surface imaging system
Serious adverse events | continuously during treatment up to 7 weeks
  mask-induced and no-mask-induced events will be recorded during treatment
Device Deficiencies of the surface guidance system | continuously during treatment up to 7 weeks
  Device Deficiencies of the surface guidance system are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Balermpas, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No